CLINICAL TRIAL: NCT05761912
Title: Application of Ultrasound Radiomics in Ultrasound Fusion Targeted Prostate Biopsy
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Minhang Central Hospital (Other)
Collaborators: Wu Jieping Medical Foundation (Other); Shanghai Municipal Commission of Health and Family Planning (Other)
Responsible Party: Principal Investigator, Chang He, Associate Clinical Professor, Shanghai Minhang Central Hospital
Other Study IDs: Prostate Radiomics-1027
Record Dates: First submitted 2022-12-18; First posted 2023-03-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer; Ultrasound; Radiomics
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultrasound fusion targeted biopsy: Prostate ultrasound had abnormal echo and radiomics analysis showed high scores
  Interventions: Diagnostic Test: Targeted biopsy
- Systematic biopsy: Patients meeting the indications for prostate biopsy

INTERVENTIONS:
Diagnostic Test: Targeted biopsy — For the high-risk targets identified by the radiomics model, perform targeted biopsy under ultrasound fusion.
  Groups: Ultrasound fusion targeted biopsy

SUMMARY:
To predict prostate cancer by ultrasound radiomics in ultrasound fusion prostate targeted biopsy.

DETAILED DESCRIPTION:
Researchers plan to develop a diagnostic and prognostic evaluation model for prostate cancer by analyzing abnormal echoes in prostate ultrasound images through radiomics. This model will be used to guide ultrasound radiomics-fusion prostate biopsy, and its accuracy will be compared with that of systematic biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥55 years old.
2. Patients had tPSA/fPSA within 1 month before biopsy.
3. Patients had any of the following indications for prostate biopsy:

   * Suspicious prostate nodules were found by digital rectal examination
   * Suspicious lesions were detected by B-ultrasound or MRI
   * PSA>10ng/ml
   * PSA 4-10ng/ml, with abnormal f/tPSA and/or PSAD values

Exclusion Criteria:

1. malignant tumors other than prostate adenocarcinoma indicated by pathology.
2. Combined with other malignant tumors (such as rectal cancer, bladder cancer, testicular cancer, etc.) that may affect the imaging findings of transrectal ultrasound or mpMRI.
3. Other conditions that would preclude needle biopsy: cachexia, decompensation of organ function, hemorrhagic diseases, local infection, etc

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged above 55 who had an indication for prostate biopsy will be screened for eligibility.
Sampling Method: Probability Sample
Enrollment: 464 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Positive rate of ultrasound radiomics fusion targeted biopsy | Up to seventh day when the pathological results were obtained after the targeted biopsy
  Positive rate of ultrasound radiomics fusion targeted biopsy
Positive rate of systematic biopsy | Up to seventh day when the pathological results were obtained after the targeted biopsy
  Positive rate of systematic biopsy
Positive rate of mpMRI cognitive fusion targeted biopsy | Up to seventh day when the pathological results were obtained after the targeted biopsy
  Positive rate of mpMRI cognitive fusion targeted biopsy
Ultrasound radiomics parameters | The 30min following the transrectal ultrasonography
  The ultrasound images are obtained by transrectal ultrasound while prostate biopsy. Then investigators use 3D-Slicer/ITK-SNAP software to draw the area of interest (ROI). "Pyradiomics" library will be used to extract the radiomics features.

SECONDARY OUTCOMES:
Gleason's score of positive tissue | Up to seventh day when the pathological results were obtained after the targeted biopsy
  Gleason's score of positive tissue from targeted prostate biopsy. Prostate cancer was graded by Gleason score (GS) ranging from 6 to 10. Tumors of GS 6 (3 + 3) are considered low grade (LG), while GS ≥7 are high grade (HG).
PI-RADS score | Within one month prior to prostate biopsy.
  Prostate Imaging Reporting and Data System (PI-RADS) score was obtained according to multiparametric magnetic resonance imaging. PI-RADS is used to standardize interpretation of prostate MRI. Each lesion is assigned a score from 1 to 5 indicating the likelihood of clinically significant cancer. PI-RADS 1: clinically significant cancer is highly unlikely to be present; PI-RADS 2: clinically significant cancer is unlikely to be present; PI-RADS 3: the presence of clinically significant cancer is equivocal; PI-RADS 4: clinically significant cancer is likely to be present; PI-RADS 5: clinically significant cancer is highly likely to be present.
Incidence of complications | Up to the first month after the targeted biopsy
  Incidence of complications associated with prostate biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Jiaqi Huang, Principal Investigator — Minhang Hospital, Fudan University
Locations (1):
- 170th Xinsong Rd, Minhang District, Shanghai, China

IPD SHARING:
Plan to Share IPD: No